CLINICAL TRIAL: NCT04696601
Title: Rapid Screening for Olfactory Disorders in Covid-19 Infection
Acronym: OLFASCAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Because of logistical problems
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 20-PP-27
Record Dates: First submitted 2020-12-23; First posted 2021-01-06 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2020-12

CONDITIONS: Olfaction Disorders; COVID-19 Testing
Keywords: Olfaction Disorders; Hyposmia; Dysosmia; Anosmia; Covid-19
MeSH Terms: conditions — Olfaction Disorders; Anosmia; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olfactory test (Experimental): The result of the olfactory test will be compared to the result of the RT-PCR test.
  Interventions: Diagnostic Test: Olfactory test

INTERVENTIONS:
Diagnostic Test: Olfactory test — The olfactory test (Olfascan) is in the form of a paper stick, previously impregnated with an odorant (non-liquid). It is placed a few centimetres from the participant's nose at the time of the test. It is a single-use test, without contact with the participant.

SUMMARY:
Loss of smell is very frequently found in Europe during Covid-19 attack. This symptom was not initially expected as part of the classic symptomatology. This loss of smell mainly concerns patients with few or no symptoms, without criteria of severity and usually treated on an outpatient basis. As a result, given the unexpected occurrence of this symptom (with less awareness in the general and medical population) and the potential risk of contamination of Covid+ and anosmic subjects (due to their less symptomatic form), it is interesting to be able to propose large-scale screening for loss of sense of smell in order to preferentially direct subjects diagnosed as anosmic towards RT-PCR-type screening. In the medium term, the loss of smell seems to persist after the infectious phase, with delayed or persistent recovery, which can lead to negative psychological repercussions.

The objective is to propose large-scale screening of the general population for loss of sense of smell during a pandemic period, in order to facilitate diagnostic orientation of the population. The diagnosis of loss of smell will be carried out using a simple olfactory test in the form of an olfactory stick to be smelled.

ELIGIBILITY:
Inclusion Criteria:

* Subject presenting himself at the covid-19 screening centre set up by the city of Nice

Exclusion Criteria:

* Presence of a sensory deficit (auditory or visual) preventing the subject from answering the questions perfectly during the olfactory test.
* Subject receiving cancer chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Olfactory test | Day 0
  Sensitivity of the olfactory test (Olfascan) for measuring anosmia, compared to the reference diagnostic test (RT-PCR analysis).

CONTACTS AND LOCATIONS:
Overall Officials: Renaud DAVID, Dr, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No